CLINICAL TRIAL: NCT03838926
Title: Tolerability Study of Trichostatin A In Subjects With Relapsed or Refractory Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VTR-297-1101
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Relapsed or Refractory Hematologic Malignancies
Keywords: Hematologic; Malignancies; Cancer; Blood
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms; Neoplasms | interventions — trichostatin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trichostatin A (Experimental)
  Interventions: Drug: Trichostatin A

INTERVENTIONS:
Drug: Trichostatin A — Intravenous Infusion

SUMMARY:
The aim of this study is to investigate the safety and tolerability of trichostatin A in individuals with relapsed or refractory hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years at the time of signing informed consent;
* Confirmed malignant hematologic disease or lymphoid malignancy that has relapsed or is refractory to standard therapy and has exhausted all available therapies;
* Presence of measurable or evaluable disease;
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2;
* Contraceptives or other approved avoidance of pregnancy measures

Exclusion Criteria:

* Allogeneic stem cell transplant recipient presenting with graft versus host disease (GVHD) either active or requiring immunosuppression;
* Concomitantly taking anti-cancer therapy (bisphosphonates are permitted);
* Undergone major surgery ≤ 2 weeks prior to starting study drug;
* Evidence of mucosal or internal bleeding;
* Impaired cardiac function or conduction defect;
* Concurrent severe and/or uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of trichostatin A measured by spontaneous reporting of adverse events (AEs) | Up to 24 months
  Measured by spontaneous reporting of adverse events (AEs)
Dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) of trichostatin A | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (4):
  - Vanda Investigational Site, Washington D.C., District of Columbia
  - Vanda Investigational Site, Lafayette, Indiana
  - Vanda Investigational Site, Hackensack, New Jersey
  - Vanda Investigational Site, Seattle, Washington
- Poland (7):
  - Vanda Investigational Site, Biała Podlaska
  - Vanda Investigational Site, Katowice
  - Vanda Investigational Site, Krakow
  - Vanda Investigational Site, Opole
  - Vanda Investigational Site, Skorzewo
  - Vanda Investigational Site, Warsaw
  - Vanda Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: No